CLINICAL TRIAL: NCT00003406
Title: A Phase I-II Intensive-Dose Ifosfamide, Carboplatin and Taxotere (IC-T) Combination Chemotherapy Followed by Autologous Stem Cell Rescue for Patients With Refractory Malignancies
Brief Title: Combination Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Refractory Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Treatment Centers of America (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066415; MRMC-CTCA-9711; NCI-V98-1446
Record Dates: First submitted 1999-11-01; First posted 2004-08-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2007-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous/Nonmalignant Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; primary systemic amyloidosis; non-Hodgkin lymphoma during pregnancy; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone | interventions — Carboplatin; Docetaxel; Ifosfamide; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel
Drug: ifosfamide
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining docetaxel, ifosfamide, and carboplatin followed by peripheral stem cell transplantation in treating patients with refractory cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the toxicities, safety, and antitumor activity of intensive high dose chemotherapy consisting of ifosfamide, carboplatin, and docetaxel followed by autologous stem cell transplantation in a variety of refractory malignancies.

OUTLINE: This is dose-escalation study of docetaxel. Cohorts of at least 4 patients each receive escalating doses of docetaxel IV over 11 hours as a continuous infusion 2 times daily in combination with constant doses of ifosfamide IV over 60 minutes daily and carboplatin IV over 60 minutes daily on days -6, -5, -4, and -3. On day 0, patients receive autologous stem cell (or bone marrow) transplantation. If 1 or 2 of 4 patients experience dose limiting toxicity (DLT), 4 additional patients are entered at the same dose level. If 3 or more of 4 or 8 patients experience DLT, there is no further dose escalation and 6 additional patients are entered at the preceding dose level. The maximum tolerated dose is defined as the dose level immediately preceding the level that caused DLT in greater than 50% of patients. Patients are followed at 3 and 6 months and then semiannually thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignancy Malignant lymphoma - Non-Hodgkin's lymphoma Intermediate and high grade (aggressive) histology with primary refractory disease or relapsed following standard therapy - Hodgkin's disease Relapsed or refractory after 2 regimens of curative therapy - No CNS disease that has not responded to standard therapy prior to bone marrow transplantation Breast cancer Stage IV disease, refractory, or relapsed after doxorubicin based first line therapy Ovarian cancer Primary refractory disease or relapsed after first line chemotherapy Testicular cancer Relapsed or refractory disease after 2 regimens of chemotherapy Other malignancies Recurrent or refractory to standard chemotherapy regimens, but with documented responses to a minimum of 2 courses of a docetaxel based chemotherapy Must not be greater than 60 days past completion of adjuvant or induction therapy Prior history of cerebrospinal fluid (CSF) tumor involvement without symptoms or signs allowed provided the CSF is now free of disease on lumbar puncture and CT scan of the brain No active leptomeningeal involvement or brain metastases No severe symptomatic CNS disease Hormone receptor status: Not specified

NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 65 and under Menopausal status: Not specified Performance status: Karnofsky 80-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT and SGPT no greater than 2.5 times normal No history of severe hepatic dysfunction Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: Ejection fraction at least 50% No major heart disease No angina pectoris No major ventricular dysrhythmias Hypertension or congestive heart failure that is controlled with medications allowed Pulmonary: DLCO at least 60% of normal No symptomatic obstructive or restrictive disease Other: HIV negative No uncompensated major thyroid or adrenal dysfunction No insulin-dependent diabetes mellitus No active infections No significant skin breakdown from tumor or other disease Must have been seen and evaluated by a dentist for teeth cleaning and potential sources of infection No other prior malignancy except nonmelanoma skin cancer Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior total dose of doxorubicin or daunorubicin of 450 mg/m2 or greater unless an endomyocardial biopsy shows less than grade 2 drug effect Endocrine therapy: Not specified Radiotherapy: No prior pelvic irradiation Surgery: Not specified Other: No concurrent nitroglycerin or antiarrhythmic drugs

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-10; Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Francisco Ballester, MD, Study Chair — Cancer Treatment Centers of America
Locations (1):
- Midwestern Regional Medical Center, Zion, Illinois, United States